CLINICAL TRIAL: NCT04749797
Title: Randomized Study Of Cranial Blocks For Postoperative Anesthesia To Reduce Pain And Postoperative Opioid Usage
Brief Title: Cranial Blocks for Postoperative Anesthesia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left institution
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Timothy Lucas, MD, PHD, MHCI, Primary Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 834603
Record Dates: First submitted 2021-01-11; First posted 2021-02-11 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Craniotomy Surgery
Keywords: craniotomy
MeSH Terms: interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of three groups: saline, bupivacaine, liposomal bupivacaine
Who Masked: Participant, Care Provider
Masking Description: On the morning of the procedure, participants will be assigned sequentially to the lowest unassigned randomization number. The surgeon performing the procedure and operating room staff will not be blinded to the intervention, since they will see whether the patient is receiving liposomal bupivacaine, bupivacaine or saline. However, all providers obtaining post-operative data from the patients will be blinded as to which treatment the patient received, in addition to the patient themselves.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Saline group (Placebo Comparator): The surgeon will administer injectable saline as a cranial block. The supraorbital, supratrochlear, zygomaticotemporal, auriculotemporal, postauricular lesser and greater occipital nerve branches on the ipsilateral side of the operation will be blocked with 5-10 cc of solution (with a maximum of 60 cc at all sites) by needle infiltration. This process generally takes 1-2 minutes. Following this, the general anesthesia is lightened and the patient is extubated in usual fashion.
  Interventions: Drug: Saline
- Bupivacaine (Active Comparator): The surgeon will administer bupivacaine as a cranial block. The supraorbital, supratrochlear, zygomaticotemporal, auriculotemporal, postauricular lesser and greater occipital nerve branches on the ipsilateral side of the operation will be blocked with 5-10 cc of solution (with a maximum of 60 cc at all sites) by needle infiltration. This process generally takes 1-2 minutes. Following this, the general anesthesia is lightened and the patient is extubated in usual fashion.
  Interventions: Drug: Bupivacaine Injection
- Liposomal Bupivacaine (Experimental): The surgeon will administer Exparel (liposomal bupivacine) as a cranial block. 20 mL of Exparel will be diluted with saline to constitute 60 mL total. The supraorbital, supratrochlear, zygomaticotemporal, auriculotemporal, postauricular lesser and greater occipital nerve branches on the ipsilateral side of the operation will be blocked with 5-10 cc of solution (with a maximum of 60 cc at all sites) by needle infiltration. This process generally takes 1-2 minutes. Following this, the general anesthesia is lightened and the patient is extubated in usual fashion.
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Used as cranial block for craniotomy surgery
  Arms: Liposomal Bupivacaine
Drug: Bupivacaine Injection — Used as cranial block for craniotomy surgery
  Arms: Bupivacaine
Drug: Saline — Used as cranial block for craniotomy surgery
  Arms: Saline group

SUMMARY:
This study compares the standard of care to the standard of care plus the administration of bupivacaine or liposomal bupivacaine in patients receiving craniotomies.

DETAILED DESCRIPTION:
Objective: To assess the effectiveness of analgesia by scalp nerve block with various agents in the first 72 hours following elective craniotomy.

The investigators will employ a randomized, single-blinded, prospective study design. Participants will be randomized 1:1:1 into one of three treatment groups: Bupivacaine, Liposomal Bupivacaine, and Saline.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Need for elective supratentorial craniotomy
* Preoperative GCS > 13

Exclusion Criteria:

* Preoperative GCS ≤ 13
* Child (<18 years of age)
* Inability to understand or use the visual analog scale (VAS)
* Proven or suspected allergy to local anesthetics
* Craniotomy incision extending beyond the field of the block
* Patients chronically (more than 2 wk) treated with narcotic medications
* Previous scalp incision
* Bilateral craniotomies
* Allergies to local anesthetics
* GCS verbal score < 4 after extubation
* Patients whose surgeries extend past 6 hours (will be placed on standard of care and removed from study)
* Patients currently on ergot-type oxytoxic drugs, MAOIs, or certain antidepressants
* Lactating Mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy H Lucas, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
No plan at this time to share data with other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saline Group | Bupivacaine | Liposomal Bupivacaine
Started | 3 | 4 | 4
Completed | 2 | 4 | 4
Not Completed | 1 | 0 | 0
Not completed — Did not meet I/E criteria after surgery | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Saline Group: The surgeon will administer injectable saline as a cranial block according to a technique previously described by Pinosky et al (Pinosky et al., 1996). The supraorbital, supratrochlear, zygomaticotemporal, auriculotemporal, postauricular lesser and greater occipital nerve branches on the ipsilateral side of the operation will be blocked with 5-10 cc of solution (with a maximum of 60 cc at all sites) by needle infiltration. This process generally takes 1-2 minutes. Following this, the general anesthesia is lightened and the patient is extubated in usual fashion.
  Saline: Used as cranial block for craniotomy surgery
- Bupivacaine: The surgeon will administer bupivacaine as a cranial block according to a technique previously described by Pinosky et al (Pinosky et al., 1996). The supraorbital, supratrochlear, zygomaticotemporal, auriculotemporal, postauricular lesser and greater occipital nerve branches on the ipsilateral side of the operation will be blocked with 5-10 cc of solution (with a maximum of 60 cc at all sites) by needle infiltration. This process generally takes 1-2 minutes. Following this, the general anesthesia is lightened and the patient is extubated in usual fashion.
  Bupivacaine Injection: Used as cranial block for craniotomy surgery
- Liposomal Bupivacaine: The surgeon will administer Exparel (liposomal bupivacine) as a cranial block according to a technique previously described by Pinosky et al (Pinosky et al., 1996). 20 mL of Exparel will be diluted with saline to constitute 60 mL total. The supraorbital, supratrochlear, zygomaticotemporal, auriculotemporal, postauricular lesser and greater occipital nerve branches on the ipsilateral side of the operation will be blocked with 5-10 cc of solution (with a maximum of 60 cc at all sites) by needle infiltration. This process generally takes 1-2 minutes. Following this, the general anesthesia is lightened and the patient is extubated in usual fashion.
  Liposomal bupivacaine: Used as cranial block for craniotomy surgery
- Total: Total of all reporting groups
Arm/Group | Saline Group | Bupivacaine | Liposomal Bupivacaine | Total
Number analyzed (Participants) | 3 | 4 | 4 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 3 | 7
  >=65 years | 1 | 2 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 1 | 2 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 2 | 4 | 4 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale
Description: The Visual Analogue Scale (VAS) is a straight, horizontal line of fixed length, numbered 0 to 10 as a measure of pain severity. The ends are the extreme limits of this scale, with the left side (0) representing the best outcome (no pain), and the right side (10) representing the worst outcome, extreme pain. The other numbers in between are representations of the variation in pain between these two feelings. The scale is presented to the participant with a verbal explanation of its meaning, and the participant points to or states a number indicating where they feel their pain level is best represented on the scale. That number is recorded.
  For each group, every participant reported several different pain scores over multiple hours. The averages (means) below represent the summation of all of the pain scores reported throughout their admission.
Time Frame: 10 months (study terminated prior to completion)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Bupivacaine | Saline Group | Liposomal Bupivacaine
Number analyzed (Participants) | 4 | 2 | 4
score on a scale | 4.5 [0 to 10] | 3 [0 to 10] | 4.25 [0 to 10]

2. Secondary Outcome: Length of Stay (ICU and
Description: The secondary outcome variables are the duration of stay in the intensive care unit (ICU), and the duration of time in the hospital until discharge.
Time Frame: 10 months (study terminated)
Measure: Mean (Full Range); unit: Days
Arm/Group | Bupivacaine | Saline Group | Liposomal Bupivacaine
Number analyzed (Participants) | 4 | 2 | 4
Days
  Hospital Stay | 4.25 [3 to 6] | 2.5 [2 to 3] | 6.5 [2 to 12]
  ICU Stay | .94 [.66 to 1.33] | .97 [0.79 to 1.16] | 1.09 [.91 to 1.33]

ADVERSE EVENTS:
Time Frame: AE data collected 72 hours post-operatively
Description: Does not differ from clinicaltrials.gov definition
Arm/Group | Saline Group | Bupivacaine | Liposomal Bupivacaine
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline Group (N=3) | Bupivacaine (N=4) | Liposomal Bupivacaine (N=4)
Edema, cerebral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 4 edema. Participant had extensive edema prior to surgery. Post-op head CT still demonstrated cerebral edema, while ultimately required further intervention, including decompressive hemicraniectomy.
Transient ischemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Subject experienced a TIA post-operatively. Symptoms resolved within the same day.

LIMITATIONS AND CAVEATS:
Study concluded before reaching subject n goal due to slow enrollment related to COVID-19 pandemic and PI leaving institution. Sample size not significant enough to accurately analyze data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT04749797/Prot_SAP_000.pdf